CLINICAL TRIAL: NCT05860907
Title: A Multicenter, Open-label, Randomized, Controlled, Prospective Clinical Study of Huaier Granules in Patients With Advanced Breast Cancer Without Visceral Metastasis
Brief Title: Clinical Study of Huaier Granules in Patients With Advanced Breast Cancer Without Visceral Metastasis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-202210-01
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer Stage IV
Keywords: non-visceral metastasis; Huaier granule; randomized controlled; prospective clinical study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaier Granule+Standard treatment (Experimental): The subject is administered according to the clinical dosage and method of medication until disease progression occurs or the subject is unable to tolerate treatment.Subjects receiving routine diagnosis and treatment simultaneously.
  Interventions: Drug: Huaier Granule
- Standard treatment (No Intervention): Subjects receive routine diagnosis and treatment without taking Huaier granules.

INTERVENTIONS:
Drug: Huaier Granule — 10g each time, three times a day
  Other Names: Z20000109（NMPA Approval Number）
  Arms: Huaier Granule+Standard treatment

SUMMARY:
This is a multicenter, open-label, randomized controlled, prospective clinical study to evaluate the efficacy and safety of Huaier Granules in patients with advanced breast cancer without visceral metastasis.

DETAILED DESCRIPTION:
This study used a blank control design and included at least 384 subjects. The experimental group and control group were randomized in a 2:1 ratio (at least 256 subjects in the experimental group and at least 128 subjects in the control group). Patients in the experimental group were treated with Huaier Granules (10g/dose, 3 times/day), while undergoing routine diagnosis and treatment; The control group received routine diagnosis and treatment, but did not take Huaier granules until the subjects experienced disease progression or intolerance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 75, regardless of gender.
* For breast cancer patients who are clinically or pathologically diagnosed as non visceral metastasis, if the patient has only local recurrence or metastasis, the clinician judges that it is not suitable or refuses to use local treatment with radical intensity, such as surgical resection or radiotherapy.
* Prior to enrollment, no more than first-line chemotherapy/endocrine therapy/targeted therapy/immunotherapy were allowed;If the patient has previously received first-line therapy, the outcome of treatment should be clinically assessed as disease progression or intolerance.
* There is at least one measurable lesion that meets the RECIST 1.1 standard, or only bone metastases (including osteolytic lesions or mixed lesions).
* The liver and kidney functions meet the following conditions: AST and ALT<3 ULN, total bilirubin ≤ 2 ULN, and blood creatinine<1.5 ULN.
* Other laboratory tests meet the following requirements: Hb ≥ 9g/dl, platelet count ≥ 60 × 10^9/L, absolute neutrophil count>1.0 × 10^9/L.
* Expected survival time ≥ 12 weeks.
* The patient's ECOG physical state score is 0 or 1.
* The subjects participated in the study voluntarily and signed an informed consent form.

Exclusion Criteria:

* Any other malignancies diagnosed within 5 years prior to enrollment, except those with a low risk of metastasis and death (5-year survival > 90%), such as adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ.
* There is visceral metastasis of breast cancer.
* Patients with advanced (local recurrence or metastasis) breast cancer who plan to receive radical local treatment.
* Serious infections (CTCAE>Level 2) have occurred within 4 weeks prior to enrollment, such as severe pneumonia, bacteremia, infection complications that require hospitalization; Symptoms and signs of infection or the need for oral or intravenous antibiotic treatment within 2 weeks prior to enrollment, except for prophylactic use of antibiotics.
* Suffering from severe acute and chronic diseases.
* Suffering from severe diabetes whose blood sugar cannot be effectively controlled.
* Patients who cannot take oral medication or are allergic to the ingredients of Huaier granules.
* Drug abusers, or those who suffer from psychological or mental illnesses that may interfere with research compliance.
* Pregnant or lactating women.
* The researcher believes that it is not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Investigator evaluated progression free survival | start of treatment until 3.5-year follow-up
  The time from randomization to the first occurrence of disease progression or death from any cause. As long as the subject experiences either "disease progression" or "death" first, it reaches the endpoint of the study

SECONDARY OUTCOMES:
Overall survival(OS) | start of treatment until 3.5-year follow-up
  The time from randomization to death (from any cause)
Clinical benefit rate (CBR) | start of treatment until 3.5-year follow-up
  The percentage of patients with advanced breast cancer who achieved a complete response, partial response, or stable disease for at least six months after treatment
Objective response rate (ORR) | start of treatment until 3.5-year follow-up
  Proportion of patients whose breast cancer has shrunk to a predetermined volume and maintains a minimum time limit
Adverse reactions | start of treatment until 3.5-year follow-up
  Harmful reactions of Huaier granules that are unrelated to the purpose of the medication under normal usage and dosage

OTHER OUTCOMES:
Reduction rate of immune-related cytokines | The baseline period，12th week±14 days and 168th week±14 days
  During the treatment process, the decrease rate of immune related cytokines（Such as IL-1 β， IL-2，IL-4，IL-5，IL-6，IL-8，IL-10，IL-12，IL-17，TNF- α， IFN- α， IFN- γ etc.） compared to the baseline period

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Professor, Principal Investigator — Fudan University
Locations (13):
- China (13):
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nantong First People's Hospital, Nantong, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The International Peace Maternity & Child Health Hospital of China welfare institute, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Hospital of Jiaxin, Jiaxin, Zhejiang
  - Lishui Municipal Central Hospital, Lishui, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No